CLINICAL TRIAL: NCT00606437
Title: Total Body Irradiation With Fludarabine Conditioning Followed by Transplantation With Combined Umbilical Cord Blood Grafts
Brief Title: Total Body Irradiation With Fludarabine Followed by Combined Umbilical Cord Blood (UCB) Transplants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00009529
Record Dates: First submitted 2008-01-07; First posted 2008-02-04 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Lymphoma; Myeloma; Leukemia; Myelodysplasia; Solid Tumors; Hodgkin's Disease; Myelofibrosis
Keywords: Umbilical Cord Blood Graft; Stem Cell Transplantation
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell; Leukemia; Anemia, Refractory, with Excess of Blasts; Hodgkin Disease; Primary Myelofibrosis | interventions — Whole-Body Irradiation; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Total Body Irradiation (TBI)/Flu Conditioning followed by combined UCB
  Interventions: Procedure: Total Body Irradiation with Fludarabine in UCB Transplants

INTERVENTIONS:
Procedure: Total Body Irradiation with Fludarabine in UCB Transplants — Administration of the preparative regimen, infusion of the stem cell graft, inpatient care during the immediate post-transplant period and outpatient follow-up for the first 3 months after transplant and at 6, 12, 24 and 36 months. Patients will have human leukocyte antigen (HLA) serologic typing and DNA typing. Bags of UCB are thawed, and diluted by 1:1 volume using a 5% albumin/dextran solution. The thawed and diluted umbilical cord blood unit (UCBU) is next weighed and centrifuged. Specimens are obtained for cell count and viability, culture, clonogenic assays, and phenotype. The UCB is infused at a rate of 1-3 ml/min. Furosemide (0.5-1.0 mg/kg/dose) may be given if volume overload or decreased urine output occurs. Each UCB infusion shall be tested for sterility, CFU content, number of CD34+ cells, cell count and viability.

SUMMARY:
Results to date of umbilical cord blood transplantation in adult and fully mature adolescent patients are inferior to what is seen in children, due to a lower stem cell dosage in adults and a more toxic conditioning regimen. This phase 1 protocol will use a potentially less toxic bone marrow conditioning regimen, followed by infusion of a combined umbilical cord blood graft that will provide the patient with a higher stem cell dose than can be given with a single umbilical cord blood infusion. The subjects will be conditioned with a total body irradiation (TBI) 13.5 Gy and fludarabine. Following conditioning, up to two unrelated, partially matched umbilical cord blood grafts will be infused that will provide a minimum nucleated cell dose of 3 x 10e7/kg . The primary objective of this study is to measure the frequency of treatment-related toxicity and engraftment.

DETAILED DESCRIPTION:
Results to date of umbilical cord blood transplantation in adult and fully mature adolescent patients are inferior to what is seen in children. There are two reasons for this. First is that the stem cell dose, measured in nucleated cells/kg body weight, is considerably lower due to the size of the recipient. This results in a higher incidence of graft failure, delayed engraftment, and impaired immune reconstitution. Multiple studies have suggested that a nucleated cell dose below 1.5 to 2 x 107/kg results in an unacceptably high risk for graft failure. Only a minority of adult patients will have a suitably matched umbilical cord blood unit that contains more than 1.5 x 107 nucleated cells/kg. The second reason for inferior outcome of umbilical cord blood transplantation in adult patients is that in comparison to children, the conventional myeloablative bone marrow conditioning regimens are more toxic. This phase 1 protocol will use a potentially less toxic bone marrow conditioning regimen, followed by infusion of a combined umbilical cord blood graft that will provide the patient with a higher stem cell dose than can be given with a single umbilical cord blood infusion. The subjects will be conditioned with a TBI 13.5 Gy and fludarabine. Fludarabine pharmacokinetics will be measured and correlated with the kinetics of donor cell engraftment as well frequency of treatment-related toxicity. Following conditioning, up to two unrelated, partially matched umbilical cord blood grafts will be infused that will provide a minimum nucleated cell dose of 3 x 10e7/kg. The primary objective of this study is to measure the frequency of treatment-related toxicity and engraftment.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 to 65 years.
* Available cord blood graft.
* Patients with high risk ALL in first complete remission, with high risk being defined by the presence of t(4;11), t(9;22) or t(1;19) or patients presenting with extreme hyperleukocytosis (WBC > 500,000/ul) or partial remission after induction therapy.
* Adult patients with acute non-lymphocytic leukemia (ANLL) in first complete remission with high-risk cytogenetics (monosomy chromosome 5 or 7, del (5q), abn (3q26), complex karyotypic abnormalities) or failure to achieve complete remission after standard induction therapy.
* All patients with ALL or ANLL in second or subsequent remission or partial remission.
* All patients with CML in chronic (failed interferon and/or Gleevec) or accelerated phase.
* Patients with myelodysplastic syndrome with International Prognostic Scoring System (IPSS) risk category of INT-1 or greater.
* Patients with severe aplastic anemia must have failed immunosuppressive therapy such as cyclosporine plus anti-thymocyte globulin.
* Non-Hodgkin's lymphoma or Hodgkin's disease:

  * High risk disease in first complete or partial remission
  * Chemotherapy-resistant relapse
  * Second or subsequent relapse or remission
* Myelofibrosis with myeloid metaplasia.
* High risk, congenital immunodeficiency disorders resulting in recurrent (> 3 episodes) life-threatening infection, known to be curable with allogeneic stem cell transplantation (to include, but not limited to; severe combined immunodeficiency disorder, combined immunodeficiency disease, Wiskott-Aldrich syndrome, Chediak-Higashi syndrome, chronic granulomatous disease, leukocyte adhesion deficiency, hemophagocytic lymphohistiocytosis).
* Patients with a history of CNS disease must have been treated and have no active CNS disease at the time of protocol treatment.
* ECOG performance status < or equal to 2.
* Patients must have adequate function of other organ systems as measured by:

  * Creatinine clearance (by Cockcroft Gault equation) > or equal to 30 ml/min. Hepatic transaminases (ALT/AST) < or equal to 4 x normal, bilirubin < or equal to 2.0 mg/dl
  * Pulmonary function tests demonstrating FVC and FEV1 of > or equal to 50% of predicted for age and DLCO > or equal to 50% of predicted
  * Ejection fraction of > or equal to 45% by echocardiogram, radionuclide scan or cardiac MRI
* Patients must be HIV negative.
* They do not have an HLA-ABC/DR identical related bone marrow or UCB donor.
* They do NOT have a 5/6 antigen matched related bone marrow or UCB donor.
* Their condition precludes waiting to search and find a donor in the National Marrow Donor Registry or an 8/8 (HLA-A, B, C, DRB1) antigen by high resolution (allele-level) typing matched unrelated donor was not found.
* Patients must not be pregnant.

Exclusion Criteria:

* Patients that have circulating antibodies specific for donor major histocompatibility antigens (as determined by panel of reactive antibody assay).
* Patients with progressive ANLL or ALL following second or third-line treatment regimens.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The primary objective will be to measure the time to and rate of hematologic engraftment following transplant and the frequency of treatment-related mortality. | 3 years

SECONDARY OUTCOMES:
The secondary objective will be to estimate the proportion of patients developing acute and chronic graft-versus-host disease, 100 day treatment-related mortality, and to measure disease-free survival. | 3 years
The tertiary objective will be to measure the time to immunologic reconstitution as defined by normal numbers of T and B cells, normal T-cell proliferative responses, normal natural killer (NK) cell function, and normal immunoglobulin synthesis. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Horwitz, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States